CLINICAL TRIAL: NCT01152619
Title: A Multi-center, Randomized, Observer-blind, Placebo-controlled Safety and Tolerability Study of Repeated Administration of Two Dose Levels of RO4989991 Administered Subcutaneously to Patients With Allergic Rhinitis
Brief Title: A Study of RO4989991 in Patients With Allergic Rhinitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP22831
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: RO4989991
- 2 (Experimental)
  Interventions: Drug: RO4989991
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Subcutaneous repeated dose
  Arms: 3; 4
Drug: RO4989991 — Subcutaneous repeated dose
  Arms: 1; 2

SUMMARY:
This multi-center, randomized, observer-blinded, placebo-controlled study will evaluate the safety and tolerability of subcutaneous doses of RO4989991 in patients with allergic rhinitis who are otherwise healthy. The anticipated time on study treatment is 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-65 years of age, inclusively
* A history of allergic rhinitis diagnosed by a physician, but otherwise healthy
* A positive skin prick test to at least one standardized allergen at screening
* A body mass index (BMI) between 18 and 32 kg/m2, inclusively

Exclusion Criteria:

* History or presence of any respiratory disease or condition other than allergic rhinitis
* Use of prescription medication or herbal remedies within 14 days of dosing the study drug
* Use of over-the-counter (OTC) medications within 7 days of dosing the study drug
* Acute infection (including viral infections) 6 weeks (8 weeks for respiratory infections) preceding dosing or any ongoing chronic infection
* Positive test for human immunodeficiency virus (HIV) or hepatitis B or C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of RO4989991 | 24 weeks

SECONDARY OUTCOMES:
Assessment of pharmacokinetics | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - South Miami, Florida
  - Normal, Illinois
  - Raleigh, North Carolina
  - Spartanburg, South Carolina